CLINICAL TRIAL: NCT03471364
Title: Double-Blinded, Placebo-Controlled Trial to Explore the Anti-Androgen, Ketoconazole, for Treating Patients With an Ongoing Epidermal Growth Factor Receptor (EGFR) Inhibitor-Induced Rash
Brief Title: Ketoconazole in Treating Participants With Ongoing EGFR Inhibitor-Induced Rash
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC17C1; NCI-2018-00355 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC17C1 (Other: Mayo Clinic in Rochester); R01CA207183 (NIH); 17-007786 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-03-06; First posted 2018-03-20 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (ketoconazole) (Experimental): Participants apply ketoconazole topically BID on days 1-28.
  Interventions: Drug: Ketoconazole; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Participants apply placebo topically BID on days 1-28.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Ketoconazole — Applied topically
  Other Names: Fungarest; Fungoral; Ketoderm; Ketoisdin; Nizoral; Orifungal M; Panfungol; R-41400; Xolegel
  Arms: Arm I (ketoconazole)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo Administration — Applied topically
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This early phase I trial studies the side effects of ketoconazole and how well it works in treating participants with ongoing EGFR inhibitor-induced rash. Ketoconazole may reduce the symptoms related to EGFR inhibitor therapy and improve EGFR inhibitor-induced rash.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate that topical ketoconazole, an anti-androgen, palliates EGFR inhibitor-induced rash within a group of racially diverse cancer patients.

II. To explore the role of ribonucleic acid (RNA) sequencing to identify other targets that might be used at a later date for rash palliation.

III. To evaluate toxicities associated with topical ketoconazole.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants apply ketoconazole topically twice daily (BID) on days 1-28.

ARM II: Participants apply placebo topically BID on days 1-28.

After completion of study treatment, participants are followed up at 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Patient has developed a rash or symptoms of a rash (cutaneous burning) characteristic of an EGFR inhibitor (health-care provider report of the rash with no other documentation is permitted)
* Patient is anticipated to continue for at least 28 days with an EGFR inhibitor or restart =< 14 days of registration and continue for at least 28 days
* Mayo only: Patient is willing to provide a skin biopsy for correlative research; Note: Can be waived with permission of study chair (documentation such as an email must be provided)
* Patient must complete baseline quality of life (QOL) packet

Exclusion Criteria:

* Patient has a prior allergy or intolerance of ketoconazole
* Patient has an allergy or intolerance to sulfites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who report an improvement in skin rash | Up to 4 weeks
  Assessed by Skindex-16. Will be estimated using the cumulative incidence function with time to improvement defined as the time from randomization to the first of the two consecutive weeks of improved symptom. The cumulative incidence of rash improvement after 4 weeks of treatment will be summarized separately by treatment arm. The difference in rash improvement incidences will be estimated and will be compared using two-sample Z-test.

SECONDARY OUTCOMES:
Incidence of skin toxicity | Up to 4 weeks
  As measured by the Skindex-16. Responses to the Skindex-16 will be categorized into three subscales: symptom, emotional, and functional. Analysis of the total scales and subscales of the Skindex-16 will involve a t-test and Wilcoxon rank sum procedures (as appropriate) at each time point as well as linear mixed modeling. Descriptive factors will be used as covariates in the modeling analysis. The change from baseline in the total score and subscales of the Skindex-16 will be compared between two arms by a two-sample, two-sided t-test. If there is evidence of non-normality (via Shapiro-Wilk testing), a non-parametric procedure such as Wilcoxon rank sum will be used.
Incidence of skin toxicity | Up to 4 weeks
  As measured by the Skin Toxicity Assessment Tool (STAT). Responses to the STAT will be categorized into three subscales: symptom, emotional, and functional. Analysis of the total scales and subscales of the STAT will involve a t-test and Wilcoxon rank sum procedures (as appropriate) at each time point as well as linear mixed modeling. Descriptive factors will be used as covariates in the modeling analysis. The change from baseline in the total score and subscales of the STAT will be compared between two arms by a two-sample, two-sided t-test. If there is evidence of non-normality (via Shapiro-Wilk testing), a non-parametric procedure such as Wilcoxon rank sum will be used.
Incidence of adverse events for ketoconazole | Up to 4 weeks
  Adverse events will be tabulated by treatment arm. Frequencies of various types of adverse events (AEs) will be compared using Fisher's exact test. Will explore the difference in reliability of the direct versus (vs.) indirect AE attribution approaches in the placebo arm.

OTHER OUTCOMES:
Change in PLA2G4D, PLOD2, and SALL4 | Baseline up to 4 weeks
  Assessed by ribonucleic acid (RNA) sequencing. Will explore the association between baseline/change in PLA2G4D, PLOD2, and SALL4 with rash improvement. Baseline gene expression level and change from baseline in gene expression level for the androgen-related genes such as PLA2G4D, PLOD2, and SALL4 will be compared between arms by t-test and Wilcoxon rank sum procedures (as appropriate). Mixed Models for Logistic Regression will also be implemented to explore the association between PLA2G4D, PLOD2, and SALL4 with rash improvement by adjusting the baseline gene expression level and change from baseline in gene expression levels for each gene. Descriptive factors will be used as covariates in the modeling analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, M.D., Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - Carle on Vermilion, Danville, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - University of Rochester, Rochester, New York

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials